CLINICAL TRIAL: NCT01489969
Title: A Double-blind, Parallel Group, Randomized, Placebo Controlled Sleep Laboratory Study of Efficacy and Safety of Neu-P11 in Insomnia Patients Aged 18-80
Brief Title: Sleep Laboratory Study to Investigate the Safety and Efficacy of Neu-P11 in Primary Insomnia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neu-P11-03-PSG
Record Dates: First submitted 2011-12-06; First posted 2011-12-12 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Primary Insomnia
Keywords: sleep latency; Sleep maintenance; Sleep fragmentation; Polysomnography
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Deprivation | interventions — N-(2-(5-methoxy-indol-3-yl)-ethyl)-4-oxo-4H-pyran-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 20 mg (Active Comparator): Neu-P11 dose of 20 mg
  Interventions: Drug: Neu-P11
- 50 mg (Active Comparator): Neu-P11 dose of 50 mg
  Interventions: Drug: Neu-P11
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Neu-P11

INTERVENTIONS:
Drug: Neu-P11 — 1 tablet daily 1-2 before bed time for 28 days of double blind treatment
  Other Names: Melatonin agonist

SUMMARY:
This is a phase II study. It is conducted using a randomized, double-blind, 3-arm placebo controlled, parallel group design. Eligible patients will be randomized in a 1:1:1 ratio to receive Neu-P11 20 mg, Neu-P11 50 mg or placebo for 4 weeks The objective of this study is to assess the efficacy of Neu-P11 (20 and 50mg) on sleep continuity parameters in insomnia patients aged 18-80 years, following the first two nights (immediate effect) and at the end of 4 weeks of double-blind treatment. The primary efficacy endpoint in this study is Latency to Persistent Sleep (LPS) measured by polysomnogram (PSG) at the first two nights of treatment (nights 15-16 of the study; mean of two consecutive nights recordings). The secondary endpoints are number of awakenings after sleep onset and the duration of wake after sleep onset measured by PSG at the first two nights of treatment (nights 15-16 of the study; mean of two consecutive nights recordings).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and aged 18-80 years (both ages included).
2. Suffering from primary insomnia according to DSM-IV criteria (307.42 primary insomnia, Appendix 25.1) (based on a Sleep History Questionnaire (SHQ) that is given to the patient at Visit Day 0, Appendix 25.1).
3. Reported subjective sleep latency of at least 30 minutes on at least three nights per week for at least one month and subjective WASO of at least 45 minutes per night on at least 3 nights per week for at least one month (based on the SHQ).
4. Subjects with habitual bed time within the range of 21:00-01:00 (inclusive), as reported by the subject during screening on Day 0.
5. If female of childbearing potential, using a reliable method of contraception during the entire study duration and for at least 3 months after study drug intake.
6. Have not been using benzodiazepine (BZD) and non-BZD hypnotics or melatoninergic drugs for the past 2 weeks or more prior to Screening.
7. Have not been using psychotropic treatments for the past 3 months or more prior to Screening.
8. Are stabilized on non-psychotropic treatments for more than 3 months prior to Screening.
9. Are willing to sign a written informed consent to participate in the study.

   • After initial screening, recruited patients will enter a 2 week placebo baseline/eligibility period.

   Patients will be admitted into a sleep lab and will continue to the double blind treatment phase if polysomnography (PSG) results meet the following criteria:
10. Mean LPS ≥30 minutes on both PSG screening nights, with neither night <15 minutes.
11. Mean total sleep time (TST) ≤390 minutes, or mean WASO ≥30 minutes on both of the 2 PSG screening nights, with neither night <15 minutes.

Exclusion Criteria:

1. According to DSM IV, subjects belonging to the following groups are excluded: 780.59 (breathing related sleep disorder); 307.45 (circadian rhythm sleep disorder); 307.47 (dyssomnia not otherwise specified); 780.xx (sleep disorder due to general medical condition)
2. Subjects suffering from insomnia secondary to other causes according to the sleep history questionnaire.
3. Subjects with sleep disorders detected during PSG inclusion/habituation night, such as sleep apnea/hypopnea and periodic leg movement syndrome (with arousal) (PLMAI>10 and/or AHI > 10 per hour).
4. Use of psychotropic treatments for the past 3 months and during the study.
5. Use of strong CYP inhibitors in the preceding 3 months and during the study
6. Use of benzodiazepines or other hypnotics during preceding two weeks (including all benzodiazepines; zopiclone, zolpidem, zaleplon, barbiturates, buspirone and hydroxyzine).
7. Alcohol intake - no more than 2 alcoholic drinks per day and any consumption less than 2 hours before study drug intake.
8. Immunosuppressive medication in the preceding 3 months and during the study
9. Severe neurological, psychiatric disorders especially psychosis, anxiety and depression
10. Intercurrent acute or chronic somatic diseases likely to interact with sleep (for example: chronic pain from any etiology, benign prostatic hypertrophy likely to require surgery in the coming six months)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Pacific Research Network, San Diego, California
  - MD Clinical, Hallandale, Florida
  - Miami research Associates, South Miami, Florida
  - Sleep Disorders Centers of Georgia, Atlanta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Community Research and Sleep Management, Crestview Hills, Kentucky
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Clinilabs, Inc., New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Neu-P11 20mg: Neu-P11 dose of 20 mg
  Neu-P11: 1 tablet daily 1-2 before bed time for 28 days of double blind treatment
- Neu-P11 50mg: Neu-P11 dose of 50 mg
  Neu-P11: 1 tablet daily 1-2 before bed time for 28 days of double blind treatment
Period: Overall Study
Arm/Group | Neu-P11 20mg | Neu-P11 50mg | Placebo
Started | 45 | 47 | 45
Completed | 40 | 43 | 44
Not Completed | 5 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neu-P11 20mg | Neu-P11 50mg | Placebo | Total
Number analyzed (Participants) | 45 | 47 | 45 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (16.16) | 47.4 (13.7) | 51.1 (14.52) | 49.6 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 33 | 97
  Male | 17 | 11 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 12 | 39
  Not Hispanic or Latino | 31 | 34 | 33 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 12 | 11 | 37
  White | 31 | 35 | 32 | 98
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Latency to Persistent Sleep
Description: The primary efficacy parameter is Latency to persistent sleep (LPS) measured by the PSG at the first two nights (immediate effect) of the double blind treatment period. LPS was summarized at baseline and after two days double-blind treatment (actual and change from baseline) for each treatment group using descriptive statistics. For each treatment group, the mean score at the end of the two days was compared, adjusting for the baselinescore. An ANCOVA model was used. Lower score indicates reduction in latency to persistent sleep and thus considered improvement
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Neu-P11 20mg | Neu-P11 50mg | Placebo
Number analyzed (Participants) | 45 | 47 | 45
minutes | -22.7 (27.39) | -39.1 (36.53) | -37.5 (38.43)

2. Other Pre Specified Outcome: Number of Awakenings (NOA)
Description: The secondary efficacy parameter is number of awakenings (NOA) measured by the PSG after 28 nights of the double blind treatment period. NOA was summarized at baseline and after 28 days double-blind treatment (actual and change from baseline) for each treatment group using descriptive statistics. For each treatment group, the mean score at the end of the 28 nights was compared, adjusting for the baseline score. An ANCOVA model was used. Lower score indicates less awakenings and thus considered improvement.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: Awekenings
Arm/Group | Neu-P11 20mg | Neu-P11 50mg | Placebo
Number analyzed (Participants) | 41 | 43 | 44
Awekenings | -3.1 (10.16) | -0.1 (10.28) | 0.5 (10.26)

3. Other Pre Specified Outcome: Duration of Wake After Sleep Onset (WASO)
Description: The secondary efficacy parameter is the duration of wake after sleep onset (WASO) measured by the PSG after 28 nights of the double blind treatment period. WASO was summarized at baseline and after 28 days double-blind treatment (actual and change from baseline) for each treatment group using descriptive statistics. For each treatment group, the mean score at the end of the 28 nights was compared, adjusting for the baseline score. An ANCOVA model was used. Lower score indicates less waking time and thus considered improvement.
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Neu-P11 20mg | Neu-P11 50mg | Placebo
Number analyzed (Participants) | 41 | 43 | 44
minutes | -28.1 (42.04) | -36.1 (64.12) | -13.3 (46.23)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Neu-P11 20mg | Neu-P11 50mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/47 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/47 | 0/45
Other Adverse Events (participants affected / at risk) | 8/45 | 3/47 | 0/45
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neu-P11 20mg (N=45) | Neu-P11 50mg (N=47) | Placebo (N=45)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days